

| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Version Number: | 3.1 |
| | Effective Date: | 25-Nov-2021 |

### Statistical Analysis Plan

### Study Title

A prospective, multicenter, Phase-IV clinical trial to assess safety of Durvalumab in Indian adult patients with locally advanced, unresectable non-small cell lung cancer (NSCLC)

| Protocol/ Study Number | : | D133HC00003 |
|---|---|---|
| Sponsor Name | : | AstraZeneca Pharma India Limited |
| Sponsor Address | : | AstraZeneca Pharma India Limited Block N1, 12th |
| Y .~ | | Floor, Manyata Embassy Business Park |
| | | Rachenahalli, Outer Ring Road, Bangalore-560045 |
| Document Version | : | 2.0 |
| Document Date : | | 15-Feb-2024 |
| Author Name (s) : | | PPD |
| Designation : | | PPO |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# Table of Contents

| | Document | ] |
|-----|-----------------------------------------------------|---|
| | 6.3 Statistical Methods for Efficacy Analysis | |
| | 6.2 Efficacy Hypothesis | |
| | 6.1.2 Secondary Endpoint | |
| | 6.1.1 Primary Endpoint | |
| 0. | Endpoints Analysis Strategy | |
| c | 5.6 Radiation Treatment | |
| | 5.5 Medical/Surgical History | |
| | 5.4 Demographic and Baseline Characteristics | |
| | 5.3 Disposition of Patients | |
| | 5.2 Decimal Point | |
| | 5.1 General Considerations | |
| 5. | Patient Characteristics and Study Conduct Summaries | |
| | Sample Size and Power Calculations | |
| | 3.2 Safety Analysis Set | |
| | 3.1 Enrolled Analysis Set | |
| 3. | Population Analysis Set | |
| | 2.5 Interim Analysis | |
| | 2.4 Blinding and Un-Blinding | |
| | 2.3 Randomization | |
| | 2.2.5 Study Plan | |
| | 2.2.4 Study Flow chart | |
| | 2.2.3 Exclusion Criteria | |
| | 2.2.2 Inclusion Criteria | |
| | 2.2.1 Study Design | |
| | 2.2 Study Description | |
| | 2.1.2 Secondary Objective | |
| | 2.1.1 Primary Objective | |
| | 2.1 Study Objective | |
| 2. | Study Objective and Design | |
| | INTRODUCTION | |
| | ST OF ABBREVIATION | |
| 110 | CT OF ADDREVIATION | _ |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

| | 6.3.1 Primary Endpoint Analysis | 13 |
|---|---|---|
| | 6.3.2 Secondary Endpoint Analysis | . 14 |
| 7. R | eferences | . 14 |
| 8. | Mock Shells | . 15 |
| Tab | es | . 15 |
| Tab | e 14.1.1.1 Patient Disposition (Enrolled Analysis Set) | 15 |
| Tab | e 14.1.1.2 Summary of Analysis Population Set (Enrolled Analysis Set) | 16 |
| Tab | e 14.1.1.3 Summary of Protocol Deviation (Enrolled Analysis Set) | 17 |
| Tab | e 14.1.2 Summary of Demographic and Baseline Characteristics (Enrolled Analysis Set) | 18 |
| Tab | e 14.1.3 Summary of Significant Medical/Surgical History (Enrolled Analysis Set) | 19 |
| Tab | e 14.1.4.1 Summary of Alcohol consumption and drug abuse (Enrolled Analysis Set) | 20 |
| Tab | e 14.1.4.2 Summary of History of Tobacco (Enrolled Analysis Set) | 21 |
| Tab | e 14.1.5.1 Summary of IP Administration (Enrolled Analysis Set) | 22 |
| Tabl | e 14.1.5.2 Summary of Study drug Administration accountability (Enrolled Analysis Set) | 23 |
| Tab | e 14.1.6 Summary of Disease Characteristics Assessment (Enrolled Analysis Set) | 24 |
| Tabl | e 14.1.7 Summary of Radiation Treatment (Enrolled Analysis Set) | 25 |
| Tab | e 14.1.8 Summary of WHO Performance Status (Safety Analysis Set) | 27 |
| Tab | e 14.2.1.1 Adverse Events (Safety Analysis Set) | 28 |
| Tabl | e 14.2.1.2 Summary of Adverse Event (Safety Analysis Set) | 29 |
| | e 14.2.1.3 Summary of Treatment Emergent Adverse Events by System Organ Class and Preferred Term (Safet<br>lysis Set) | • |
| | e 14.2.1.4 Summary of Serious Treatment Emergent Adverse Events by System Organ Class and Preferred Terrety Analysis Set) | |
| | e 14.2.1.5 Summary of Treatment Emergent Adverse Events leading to permanent discontinuation by System an Class and Preferred Term (Safety Analysis Set) | |
| | e 14.2.1.6 Summary of Treatment Emergent Adverse Events leading to Death by System Organ Class and<br>erred Term (Safety Analysis Set) | . 33 |
| | e 14.2.1.7 Summary of Treatment Emergent Adverse by System Organ Class, Preferred Term and Severity (Saf<br>lysis Set) | |
| | e 14.2.1.8 Summary of Treatment Emergent Adverse by System Organ Class, Preferred Term and Relationship<br>Study Drug (Safety Analysis Set) | |
| | e 14.2.1.9 Summary of Serious Treatment Emergent Adverse by System Organ Class, Preferred Term and tionship with Study Drug (Safety Analysis Set) | 35 |
| | e 14.2.1.10 Summary of Treatment Emergent Adverse by System Organ Class, Preferred Term and Relationshin Study Drug (Safety Analysis Set) | |
| with | Study Drug (Safety Analysis Set) | 3 |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

| Table 14.3.1 Summary of Physical Examination (Safety Analysis Set) | 37 |
|---|---|
| Table 14.3.2 Summary of Vital Sign (Safety Analysis Set) | 39 |
| Table 14.3.3 Summary of 12-Lead Electrocardiogram (Safety Analysis Set) | 41 |
| Table 14.3.4.1 Summary of Haematology (Safety Analysis Set) | 43 |
| Table 14.3.4.2 Summary of Serum Chemistry (Safety Analysis Set) | 45 |
| Table 14.3.4.3 Summary of Urine Routine and Microscopy (Safety Analysis Set) | 48 |
| Table 14.3.4.4 Summary of Thyroid function test (Safety Analysis Set) | 50 |
| Table 14.3.5 Summary of Urine Pregnancy Test (Safety Analysis Set - Female) | 50 |
| Listings | 52 |
| Listing 16.1.1.1. Listing of Patient Informed Consent Details | 52 |
| Listing 16.1.1.2 Listing of Patient Eligibility Criteria and Analysis Population Set | 53 |
| Listing 16.1.1.3 Listing of Patient Study Completion / Discontinuation | 53 |
| Listing 16.1.1.4 Listing of Patient Protocol Deviation | 54 |
| Listing 16.1.2 Listing of Patient Demographics Data | 55 |
| Listing 16.1.3 Listing of Patient Medical / Surgical History | 56 |
| Listing 16.1.4.1 Listing of Patient IP Administration I | 57 |
| Listing 16.1.4.2 Listing of Patient IP Administration II | 58 |
| Listing 16.1.4.3. Listing of Patient Study Drug Administration Accountability | 59 |
| Listing 16.1.5 Listing of Patient Disease characteristics Assessment | 60 |
| Listing 16.1.6.1 Listing of Patient Alcohol consumption and drug abuse | 61 |
| Listing 16.1.6.2 Listing of Patient History of Tobacco | 62 |
| Listing 16.1.7 Listing of Patient Urine Pregnancy Test | 63 |
| Listing 16.1.8 Listing of Patient Prior/Concomitant Medications | 64 |
| Listing 16.1.9.1 Listing of Patient Radiation Treatment | 65 |
| Listing 16.1.9.2 Listing of Patient Radiation Treatment | 66 |
| Listing 16.1.10 Listing of Patient WHO Performance status | 67 |
| Listing 16.3.1.1 Listing of Patient Adverse Event | 68 |
| Listing 16.3.1.2 Listing of Patient Adverse Event | 69 |
| Listing 16.3.1.3 Listing of Patient Adverse Event | 70 |
| Listing 16.3.2 Listing of Patient Physical Examination | 71 |
| Listing 16.3.3 Listing of Patient Vital Signs | 72 |
| Listing 16.3.4 Listing of Patient 12-Lead electrocardiogram | 73 |
| Listing 16.3.5.1 Listing of Patient Haematology Parameters | |
| Description and Confidential Description | Dags 4 of 77 |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

| Listing 16.3.5.2 Listing of Patient Serum Chemistry Parameters | 75 |
|---|---|
| Listing 16.3.5.3 Listing of Patient Urine Routine and Microscopy Parameters | 76 |
| Listing 16.3.5.4 Listing of Patient Thyroid Function Tests | 77 |

# LIST OF ABBREVIATION

| Abbreviation | Term |
|------------------------------------|------------------|
| Docum | ent |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

| AE | Adverse Event |
|---|---|
| CRF | case report form (electronic/paper) |
| CSA | clinical study agreement |
| CSR | clinical study report |
| CTCAE | Common Terminology Criteria for Adverse Event |
| DAE | discontinuation of investigational product due to Adverse Event |
| DNA | deoxyribonucleic acid |
| EC | ethics committee, synonymous to institutional review board (IRB) |
| | and independent ethics committee (IEC) |
| GCP | Good Clinical Practice |
| ICH | International Conference on Harmonisation |
| International Co-ordinating | If a study is conducted in several countries the International Co- |
| investigator | ordinating Investigator is the Investigator co-ordinating the |
| | investigators and/or activities internationally. |
| IVRS | interactive voice response system |
| IWRS | interactive web response system |
| LSLV | last subject last visit |
| LIMS | laboratory information management system |
| OAE | other significant Adverse Event |
| PI | principal investigator |
| SAE | serious Adverse Event |
| SAP | statistical analysis plan |
| WBDC | web based data capture |

# 1. INTRODUCTION

The purpose of this document is to provide a description of the statistical methods and procedures to be implemented for the analysis of data from D133HC00003 study. This document is based on protocol version 4.1 Dated 12-Oct-2022.



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

The statistical planning and conduct of analysis of the data from this study will follow the principles defined in relevant ICH-E9 guidelines. Any change from the planned analysis as described in the protocol, are detailed here, and any differences described here supersede the analysis as presented in the protocol.

# 2. Study Objective and Design

### 2.1 Study Objective

#### 2.1.1 Primary Objective

To assess the safety of durvalumab among locally advanced unresectable non-small cell lung carcinoma in Indian patients

#### 2.1.2 Secondary Objective

Not Applicable

#### 2.2 Study Description

#### 2.2.1 Study Design

This is a Phase IV, open-label, single arm, multi-center, prospective study to be conducted in India. Two cohorts of patients will be included in the current study patients with locally advanced, unresectable NSCLC whose disease has not progressed following platinum-based chemoradiation therapy (N= 100). Potential patients will undergo eligibility determination within 7 days prior to first dose. Patients who meet the protocol-defined inclusion/exclusion criteria will be prospectively enrolled in a sequential manner at 10 centres in India. All enrolled patients will be treated with durvalumab administered intravenously over 60 minutes at 10 mg/kg every 2 weeks. The treatment period for this study is 20 weeks, which corresponds to 10 doses of study drug administration. Treatment will continue as long as clinical benefit is observed for a maximum of 20 weeks or either of the criteria defined in section 7 are met, whichever is earlier. Patients who are observed to continue to receive clinical benefit from durvalumab at end of Week 20 will continue treatment in post-trial phase. Any patient who discontinues treatment with durvalumab before end of Week 20 on study will be followed for 90 days after discontinuation of study drug or until the start of alternate treatment intervention, whichever is earlier. Safety will be evaluated throughout the evaluation phase and during the follow up of patients who discontinue treatment before end of Week 20 by physical exams including vital signs, AE/SAE monitoring, laboratory evaluations and recording of concomitant medications.



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

#### 2.2.2 Inclusion Criteria

Patients are eligible to be included in the study only if all of the following inclusion criteria and none of the exclusion criteria apply:

- 1. Provision of signed, written and dated informed consent prior to any study specific Procedures
- 2. Male or female aged 18 years or older
- 3. As per local prescribing information and in view of positive benefit-risk assessment, patient prescribed Durvalumab treatment as per independent clinical judgment of treating physician for either treatment for locally advanced, unresectable non-small cell lung carcinoma whose disease has not progressed following platinum-based chemoradiation therapy (N= 100)

#### 2.2.3 Exclusion Criteria

- Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study
  or the follow-up period of an interventional study
- 2. Current or prior use of immunosuppressive medication within 14 days before the first dose of study drug, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. Systemic steroid administration required to manage toxicities arising from radiation therapy delivered as part of the chemoradiation therapy for locally advanced NSCLC is allowed.
- 3. Prior exposure to any anti-PD-1 or anti-PD-L1 antibody including durvalumab.
- 4. For NSCLC cohort only:
  - a. Mixed small cell and non-small cell lung cancer histology
  - b. Any unresolved toxicity CTCAE > Grade 2 from the prior chemoradiation therapy.
  - c. Patients with ≥Grade 2 pneumonitis from prior chemoradiation therapy
- Active or prior documented autoimmune disease within the past 2 years, inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis), primary immunodeficiency, organ transplant that requires therapeutic immunosuppression, hypersensitivity to study drug or any excipient, leptomeningeal carcinomatosis, tuberculosis.
  - NOTE: Patients with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
- Female patients who are pregnant, breast-feeding or male or female patients of reproductive potential who
  are not employing an effective method of birth control



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Any condition that, in the opinion of the investigator, would interfere with evaluation of the study drug or interpretation of patient safety or study results.

# 2.2.4 Study Flow chart





| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# 2.2.5 Study Plan

| Dose | | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Days (± 3 days of windows period) | -7 to 0 | 1 | 15 | 29 | 43 | 57 | 71 | 85 | 99 | 113 | 127 | 141 | 230 |
| Week (1st day of week) | | 0 | 2 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 18 | Last day of<br>week 20 | |
| Visit | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | ll | 12 | 13 |
| | Screening<br>Period | Evaluation Phase | | | | | | Follow-up<br>period | | | | | |
| | Screening<br>Visit | | | | Ev | aluatio | n Visi | (2-11) | ) | | | End of<br>Evaluation<br>Visit | End of Study<br>Visit |
| Informed Consent Form | X | | | | | | | | | | | | |
| Eligibility Criteria | X | X | | | | | | | | | | | |
| Demography and history of tobacco and alcohol use | X | | | | | | | | | | | | |
| Medical and surgical history (including all<br>treatments for NSCLC/mUC) | X | | | | | | | | | 1 | | | |
| Physical examination | X | X Targeted physical exam (based on symptoms) X | | | | X | | | | | | | |
| Vital signs (pre and post-infusion vital signs assessments; see Section 6.4.8) | | X | X | X | X | X | X | X | X | X | X | X | |
| Urine Pregnancy Test | X | | | | | | | | | | | | |
| Weight | | X | | X | | X | | X | | X | | | |
| World Health Organization performance status | X | X | X | X | X | X | X | X | X | X | X | X | |
| Concomitant medications | X | X | X | X | X | X | X | X | X | X | X | X | |
| Disease Characteristics Assessment | | X | | | X | | | X | | | X | X | |
| Adverse event/serious adverse event assessment | | X | X | X | X | X | X | X | X | X | X | X | X |
| Electrocardiogram (before dosing of IP) | | X | | | | X | | | | X | | | |
| Haematology | | X | X | X | X | X | X | X | X | X | X | X | |
| Serum chemistry (LFT, RFT, Electrolytes) | | X | X | X | X | X | X | X | X | X | X | X | |
| Urine Routine and microscopy | | X | X | X | X | X | X | X | X | X | X | X | |
| Thyroid function tests (TSH, T3 and T4) <sup>a</sup> | | X | | | | X | | | | X | | X | |
| IP Administration | | X | X | X | X | X | X | X | X | X | X | | |

a. Except screening visit, free T3 and free T4 will only be measured if TSH is abnormal or if there is clinical suspicion of an AE related to the endocrine system.

| Proprietary | and | Confide | ntial | Document |
|-------------|-----|---------|-------|----------|



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

#### 2.3 Randomization

Not Applicable

### 2.4 Blinding and Un-Blinding

Not Applicable

#### 2.5 Interim Analysis

No interim analyses is planned for this study.

### 3. Population Analysis Set

### 3.1 Enrolled Analysis Set

The enrolled population is defined as all screened patients who provided written informed consent at screening assessment, satisfied all the eligibility criteria and enrolled into the study.

### 3.2 Safety Analysis Set

All the patients who are enrolled into the study and received at least one dose of investigational product as an IV infusion.

# 4. Sample Size and Power Calculations

The primary endpoint of the trial is to demonstrate the safety profile of durvalumab in routine clinical practice as assessed by the incidence of Adverse Events (AEs) (Serious and Non-serious AEs) observed during trial. Based on the Durvalumab historic data, estimated proportion of 31% for Adverse Events prevalence rate. With a sample size of 83, would be able to achieve the 10% precision of the estimates with the 95% level of confidence. Approximately 120 participants will be screened to achieve around 100 participants enrolled in the study.

| Scenario# | estimated proportion | Precision | Confidence level | Required sample size |
|---|---|---|---|---|
| 1 | 31% | .15 | 95% | 37 |
| 2 | 31% | .14 | 95% | 42 |
| 3 | 31% | .13 | 95% | 49 |
| 4 | 31% | .12 | 95% | 58 |
| 5 | 31% | .11 | 95% | 68 |
| 6 | 31% | .10 | 95% | 83 |

| Document |
|---------------------------------------|



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# 5. Patient Characteristics and Study Conduct Summaries

#### 5.1 General Considerations

Statistical Analysis will be performed using SAS (version 9.4 or higher) software (SAS Institute Inc USA). Categorical variables will be summarized with the frequency, percentage of Patients in each category. Continuous variables will be summarized descriptively with the number of Patients, mean, standard deviation, median, minimum and maximum values.

#### 5.2 Decimal Point

Unless otherwise noted, means, median, will be presented to one decimal place more than the measured value, the same decimal as the measured value, percentages and 95% confidence intervals will be presented to two decimal places and p-value will be presented to three decimal place. Percentages after zero counts will not be displayed and percentages equating to 100% will be presented as 100%, without any decimal places.

#### 5.3 Disposition of Patients

Patient disposition table will be based on all Enrolled Analysis Set who consented to participate in the study. The following summaries will be included in the disposition table: total number of Patient Enrolled in the study, total number of Patients screened in the study, number of Patients who failed screening, number and percentage of Patients who completed the study and number and percentage of Patients who discontinued from the study with reason for discontinuation.

### 5.4 Demographic and Baseline Characteristics

Demographic and baseline characteristics will be summarized based on the Enrolled Analysis Set.

Descriptive summaries will be provided for the demographic and baseline characteristics. Demographic characteristics and baseline characteristics such as age, Gender and Weight, etc. will be summarized and tabulated for Enrolled Analysis Set.

All the continuous variables will be summarized by n, mean, standard deviation, median, minimum and maximum values. All the categorical variables will be summarized as frequency, percentage of Patients.

#### 5.5 Medical/Surgical History

Medical History will be summarized based on the Enrolled Population.

Descriptive summaries will be provided for the Medical/Surgical History.

All the continuous variables will be summarized by n, mean, standard deviation, minimum, median and maximum values. All the categorical variables will be summarized as frequency, percentage of Patients.



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

#### 5.6 Radiation Treatment

Radiation Treatment will be summarized based on the Enrolled Population.

Descriptive summaries will be provided for the Radiation Treatment.

All the continuous variables will be summarized by n, mean, standard deviation, minimum, median and maximum values. All the categorical variables will be summarized as frequency, percentage of Patients.

### 6. Endpoints Analysis Strategy

### 6.1 Endpoints Analysis

### 6.1.1 Primary Endpoint

Adverse Events (AEs), Serious Adverse Events (SAEs), and AEs of Special Interest (AESI) including interstitial lung disease/pneumonitis-like events, and on-study deaths.

### 6.1.2 Secondary Endpoint

Not Applicable

### 6.2 Efficacy Hypothesis

There is no statistical hypothesis to be tested in this study.

### 6.3 Statistical Methods for Efficacy Analysis

Statistical Analysis will be performed using SAS (version 9.4 or higher) software (SAS Institute Inc USA). Categorical variables will be summarized with the frequency and percentage of Patients in each category. Continuous variables will be summarized descriptively with the number of Patients, mean, standard deviation, minimum, median and maximum values.

### 6.3.1 Primary Endpoint Analysis

The primary analysis for primary endpoint will be based on Safety Analysis Set.

Primary Endpoint evaluations will include Adverse Events (AEs), Serious Adverse Events (SAEs), Adverse Events of Special Interest (AESI) including interstitial lung disease/pneumonitis-like events and on study Deaths.

Adverse Events (AEs), Serious Adverse Events (SAEs), Adverse Events of Special Interest (AESI) including interstitial lung disease/pneumonitis-like events and on study Deaths will be summarized using Frequency, Percentages.

Physical Examination will include General Appearance, Respiratory system, Cardiovascular system, Abdomen, Skin, Heent, Neck, Lymph node, Thyroid, Musculo-skeletal system, Genital/Rectal and Neurological System. Physical Examination will be summarized based on the Safety Analysis Set.

Descriptive summaries will be provided for the Physical Examination.



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

All the continuous variables will be summarized by n, mean, standard deviation, minimum, median and maximum values. All the categorical variables will be summarized as frequency, percentage.

Vital Signs will include Pulse rate, Respiratory rate, Systolic Blood Pressure, Diastolic Blood Pressure, Oxygen Saturation and Temperature. Vital Signs will be summarized based on the Safety Analysis Set.

Vital Signs will be summarised by number of observations, arithmetic mean, SD, median, minimum and maximum values.

12-Lead Electrocardiogram will include Heart rate, QRS, PR, RR, QT and QTcF. 12-Lead Electrocardiogram will be summarized based on the Safety Analysis Set.

12-Lead Electrocardiogram will be summarised by number of observations, arithmetic mean, SD, median, minimum and maximum values.

### 6.3.2 Secondary Endpoint Analysis

### Not applicable

#### 7. References

- AstraZeneca Pharma India Limited Block N1, 12th Floor, Manyata Embassy Business Park Rachenahalli, Outer Ring Road, Bangalore-560045.
- ICH E3 Guideline
- ICH E9; STATISTICAL PRINCIPLES FOR CLINICAL TRIALS



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# 8. Mock Shells

# Tables

Table 14.1.1.1 Patient Disposition (Enrolled Analysis Set)

| | Durvalumab<br>n (%) |
|---|---|
| | 11 (70) |
| Number of Patients Screened [1], n | xxx |
| Number of Screen failure Patients [2], n | xx |
| Number of Subjects Eligibility Criteria met | xxx |
| Number of Subjects Withdrawal/Discontinued before Study Enrolment | xx |
| Reason: | |
| XXXXXXXXX | xx |
| Xxxxx xxxxxxx | xx |
| Number of Patient Enrolled into the Study | xxx |
| Number of Patients Completed the study | xx (xx.xx) |
| Number of Patients Discontinued from the study | xx (xx.xx) |
| Reason for Discontinuation: | |
| Patient Decision | xx (xx.xx) |
| Adverse Event | xx (xx.xx) |
| Severe non-compliance to study protocol that, in the opinion of the investigator or sponsor, warrants | |
| withdrawal | xx (xx.xx) |
| Any AE that meets criteria for discontinuation | xx (xx.xx) |
| An AE related to study drug that is ≥Grade 3, with the exception of toxicities that do not meet criteria for | or |
| discontinuation | xx (xx.xx) |
| ≥Grade 3 infusion reaction | xx (xx.xx) |
| Initiation of alternative anticancer therapy including another investigational agent | xx (xx.xx) |
| Disease progression as per investigator's clinical and imaging assessment | xx (xx.xx) |
| Pregnancy or intent to become pregnant | xx (xx.xx) |
| Use of prohibited concomitant medication | xx (xx.xx) |
| Study terminated by sponsor | xx (xx.xx) |
| Death | xx (xx.xx) |
| Clinically significant abnormal laboratory value(s) | xx (xx.xx) |
| Other | xx (xx.xx) |
| XXXXXX | xx (xx.xx) |
| XXXXXX | xx (xx.xx) |

- [1] Patients who provided informed consent; [2] patients who did not satisfied the eligibility criteria i.e., Inclusion or exclusion criteria.
- The small "n" in summary statistics represents the number of patients in the row category.
- Percentages in are based on the number of patients enrolled into the study.
- Source: Listing 16.1.1.1 and Listing 16.1.1.
- Table Name: xxxxxxxx



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# Table 14.1.1.2 Summary of Analysis Population Set (Enrolled Analysis Set)

| | Durvalumab<br>N = xxx<br>n (%) |
|-----------------------|--------------------------------|
| Enrolled Analysis Set | xx (xx.xx) |
| Safety Analysis Set | xx (xx.xx) |

- The Capital "N" in the column header represents the total number of patients in Enrolled Analysis Set.
- The small "n" in summary statistics represents the total number of patients in the row category.
- Percentages are based on the total number patients in Enrolled Analysis Set.
- Enrolled Analysis Set: The enrolled population is defined as all screened patients who provided written informed consent at screening assessment, satisfied all the eligibility criteria and enrolled into the study.
- Safety Population: All the patients who are enrolled into the study and received at least one dose of investigational product as an IV infusion.

Source: Listing 16.1.1.4
 Table Name: xxxxxxxx



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.1.1.3 Summary of Protocol Deviation (Enrolled Analysis Set)

| | Durvalumab |
|------------------------------------------|------------|
| | N = xxx |
| | n (%) |
| Patient undergone any Protocol Deviation | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| Protocol Deviation | |
| Restrictions | xx (xx.xx) |
| Enrolment/IE Criteria | xx (xx.xx) |
| Out of visit window | xx (xx.xx) |
| IP Administration | xx (xx.xx) |
| Drug accountability | xx (xx.xx) |
| Noncompliance | xx (xx.xx) |
| Use of prohibited medication | xx (xx.xx) |
| Safety assessment | xx (xx.xx) |
| Other | xx (xx.xx) |
| Other 1 | xx (xx.xx) |
| Other n | xx (xx.xx) |
| Action Taken | |
| Patient continued in the study | xx (xx.xx) |
| Patient Discontinued in the study | xx (xx.xx) |
| Retraining | xx (xx.xx) |
| Other | xx (xx.xx) |
| Other 1 | xx (xx.xx) |
| Other n | xx (xx.xx) |

- The Capital "N" in the column header represents the total number of patients in Enrolled Analysis Set.
- The small "n" represents the total number of patients in the row category.
- Percentages are based on number of patients in Enrolled Analysis Set.
- Patients may have more than one protocol deviation.
- Source: Listing 16.1.1.3



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.1.2 Summary of Demographic and Baseline Characteristics (Enrolled Analysis Set)

| Demographic and Baseline Variables | N = xx |
|------------------------------------|----------------|
| Age (Years) | |
| n | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |
| Gender, n (%) | |
| Male | xx (xx.xx) |
| Female | xx (xx.xx) |
| Missing | xx (xx.xx) |
| Height (cm) | |
| N | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |
| Weight (Kg) | |
| n | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |
| Race, n (%) | |
| Indian | xx (xx.xx) |
| Other | xx (xx.xx) |
| Other 1 | xx (xx.xx) |
| Other n | xx (xx.xx) |

- The Capital "N" in the column header represents the total number of patients in Enrolled Analysis Set.
- The small "n" in summary statistics represents the total number of patients.
- Percentages are based on number of patients in Enrolled Analysis Set.
- SD = Standard Deviation, min=minimum, max=maximum
- Source: Listing 16.1.2



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.1.3 Summary of Significant Medical/Surgical History (Enrolled Analysis Set)

| System Organ Class Preferred Term | Durvalumab<br>N = xx<br>n (%) |
|---|---|
| Number of patient with at least one medical/Surgical history | xx (xx.xx) |
| System Organ Class 1 | xx (xx.xx) |
| Preferred Term 1 | xx (xx.xx) |
| Preferred Term 2 | xx (xx.xx) |
| System Organ Class 2 | xx (xx.xx) |
| Preferred Term 1 | xx (xx.xx) |
| Preferred Term 2 | xx (xx.xx) |
| System Organ Class 3 | xx (xx.xx) |
| Preferred Term 1 | xx (xx.xx) |
| Preferred Term 2 | xx (xx.xx) |

- The Capital "N" in the column header represents the total number of patients in Enrolled Analysis Set.
- The small "n" in summary statistic represents the total number of patients in the row category.
- Percentages are based on number of patients in Enrolled Analysis Set.
- System Organ Class and Preferred term are coded using standards of MedDRA version xx.x
- Patient having a medical history of similar SOC/PT more than once will be counted only once.
- Source: Listing 16.1.3
- Table Name: xxxx
- Programmer's Note 1: The above table will be continued for all other SOC and PT terms.
- Programmers Note 2: SOC and PT will be sorted in descending order of frequency.



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.1.4.1 Summary of Alcohol consumption and drug abuse (Enrolled Analysis Set)

| | Durvalumab<br>N = xx |
|---|---|
| | n (%) |
| lumber of patients with significant history of alcoholism or drug abuse | xx (xx.xx) |
| Alcohol | |
| Current | xx (xx.xx) |
| Past | xx (xx.xx) |
| Never | xx (xx.xx) |
| Drug | |
| Current | xx (xx.xx) |
| Past | xx (xx.xx) |
| Never | xx (xx.xx) |

- The Capital "N" in the column header represents the total number of patients in Enrolled Analysis Set.
- The small "n" in summary statistic represents the total number of patients in the row category.
- =Percentages are based on total number of patients in Enrolled Analysis Set.
- Source: Listing 16.1.6.1
- Table number: xxxxx



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Dlan | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

# Table 14.1.4.2 Summary of History of Tobacco (Enrolled Analysis Set)

| | Durvalumab |
|-----------------|------------|
| | N = xxx |
| | n (%) |
| Smoking History | |
| Current | xx (xx.xx) |
| Past | xx (xx.xx) |
| Never | xx (xx.xx) |

- The Capital "N" in the column header represents the total number of patients in Enrolled Analysis Set.
- The small "n" in summary statistic represents the total number of patients in the row category.
- Percentages are based on total number of patients in Enrolled Analysis Set.
- Source: Listing 16.1.6.2
- Table Name: xxxxx



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Dlan | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Table 14.1.5.1 Summary of IP Administration (Enrolled Analysis Set)

| | Durvalumab |
|-----------------------------------------|----------------|
| | N = xx |
| Visit 2 | |
| Total Dose Administered(mg/mL) | |
| n | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |
| Dose interrupted during infusion, n (%) | |
| No | xx (xx.xx) |
| Yes | xx (xx.xx) |
| Dose Restarted, n (%) | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |

- The Capital "N" in the column header represents the total number of patients in Enrolled Analysis Set.
- The small "n" in summary statistic represents the total number of patients in the row category.
- Percentages are based on number of patients in Enrolled Analysis Set.
- SD = Standard Deviation, min=minimum, max=maximum
- Source: Listing 16.1.4.1 and Listing 16.1.4.2
- Table Name: xxxxx
- Programmer Note: Continue the above table from Visit 2 to Visit 11.



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.1.5.2 Summary of Study drug Administration accountability (Enrolled Analysis Set)

| | N = xx |
|--------------------------------------------------------|----------------|
| At Visit 11, | |
| Dose Reduced in any of the Visit , n (%) | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| Dosing Completed, n (%) | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| Number of IV Dose administered in the treatment period | |
| n | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |
| Unused IP returned, n (%) | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| Compliance (%) | |
| n | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |

- The Capital "N" in the column header represents the total number of patients in Enrolled Analysis Set.
- The small "n" represents the total number of patients in the row category.
- All Percentages rows are based on number of patients in Enrolled Analysis Set.
- SD = Standard Deviation, min=minimum, max=maximum
- Source: Listing 16.1.4.3
- Table Name: xxxxx



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Dlan | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Table 14.1.6 Summary of Disease Characteristics Assessment (Enrolled Analysis Set)

| | Durvalumab |
|------------------------|------------|
| | N = xx |
| | n (%) |
| At Visit x | |
| Disease Stage of NSCLC | |
| Stage IIIA | xx (xx.xx) |
| Stage IIIB | xx (xx.xx) |
| Stage IIIC | xx (xx.xx) |

- The Capital "N" in the column header represents the total number of patients in Enrolled Analysis Set.
- The small "n" in summary statistic represents the total number of patients in the row category.
- Percentages are based on total number of patients in Enrolled Analysis Set.
- Programmer Note:- Visit x : Visit 2, Visit 5, Visit 8, Visit 11 and Visit 12.
- Source: Listing 16.1.5
- Table Name: xxxx



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Diam | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Table 14.1.7 Summary of Radiation Treatment (Enrolled Analysis Set)

| | N = xx |
|---|---|
| Clinical Stage of NSCLC | |
| Stage IIIA | xx (xx.xx) |
| Stage IIIB | xx (xx.xx) |
| Stage IIIC | xx (xx.xx) |
| Pathological staging of NSCLC done | |
| No | xx (xx.xx) |
| Yes | xx (xx.xx) |
| Stage IIIA | xx (xx.xx) |
| Stage IIIB | xx (xx.xx) |
| Stage IIIC | xx (xx.xx) |
| Histology of Tumor | |
| Squamous | xx (xx.xx) |
| Non-squamous | xx (xx.xx) |
| Technique of Radiation | |
| Sequential Communication Commu | |
| IMRT . | xx (xx.xx) |
| IGRT CONTROL OF THE PROPERTY O | xx (xx.xx) |
| Proton | xx (xx.xx) |
| SBRT | xx (xx.xx) |
| Other Other | xx (xx.xx) |
| Other 1 | xx (xx.xx) |
| Other 2 | xx (xx.xx) |
| Concurrent | |
| IMRT | xx (xx.xx) |
| IGRT | xx (xx.xx) |
| Proton | xx (xx.xx) |
| SBRT | xx (xx.xx) |
| Other | xx (xx.xx) |
| Other 1 | xx (xx.xx) |
| Other 2 | xx (xx.xx) |
| Dose of Radiation (Gy) | |
| n | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | XX.X |
| (min, max) | (xx.xx, xx.xx) |
| nduction chemotherapy given | , , |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| If Yes, Number of cycles | , -7 |
| n | Xx |

** Document** 




| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

| Mean (SD) XX.X (XX.XXX) Median (min, max) (XX.X (XX.XXX) Type of Chemotherapy Sequential Concurrent XX Number of cycles (Sequential) XX n XX Missing XX Median (SD) XX.X (XX.XXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | |
|---|---|---|
| (min, max) (xxxxx, xxxxxx) Type of Chemotherapy Sequential Concurrent Xx Number of cycles (Sequential) Xx n Xx Mean (SD) xxxx (xxxxx) Median (xxxxx) (min, max) (xxxxx, xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | Mean (SD) | xx.x (xx.xx) |
| Type of Chemotherapy Sequential Concurrent Number of cycles (Sequential) Xx n Xx Missing Xx Mean (SD) xx.x Median (xx.xx) Number of cycles (Concurrent) Xx n Xx Missing Xx Mean (SD) xx.x Median xx.x xx.x xx.x Median xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x <td>Median</td> <td>xx.x</td> | Median | xx.x |
| Sequential Concurrent Number of cycles (Sequential) n Xx Missing Xx Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) Number of cycles (Concurrent) Xx n Xx Mesning Xx Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) Mean (SD) xx.x (xx.xxx) Median xx.x (min, max) (xx.xx, xx.xxx) Performance status at time of initiation of CRT xx n Xx Missing Xx Mean (SD) xx.x (xx.xxxx) Median xx.x (xin, max) xx.x (xx.xxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | (min, max) | (xx.xx, xx.xx) |
| Concurrent Number of cycles (Sequential) n Xx Missing Xx Mean (SD) XX. (XX.XX) Median XX.X (min, max) (XX.XX) Number of cycles (Concurrent) XX n XX Missing XX Median XX.X (min, max) (XX.XX) Tumor response assessment done on imaging (days) XX n XX Missing XX Median XX.X (min, max) (XX.XXX) Performance status at time of initiation of CRT XX n XX Missing XX Missing XX Missing XX Mean (SD) XX Median XX | Type of Chemotherapy | |
| Number of cycles (Sequential) Xx n Xx Missing Xx Mean (SD) XX.X (XX.XX) Median XX.X (min, max) (XX.XX, XX.XX) Number of cycles (Concurrent) XX n XX Missing XX Median XX.X (min, max) (XX.XX, XX.XX) Tumor response assessment done on imaging (days) XX n XX Missing XX Median XX.X (min, max) (XX.XX, XX.XX) Performance status at time of initiation of CRT XX n XX Missing XX Mean (SD) XX.X Mean (SD) XX.X Mean (SD) XX.X Median XX.X Median XX.X Median XX.X (min, max) (XX.XX, XX.XX) | Sequential | |
| n Xx Missing Xx Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) Number of cycles (Concurrent) Xx n Xx Missing Xx Mean (SD) xx.x (xx.xx) Median (xx.xx, xx.xx) Tumor response assessment done on imaging (days) Xx n Xx Missing Xx Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) Performance status at time of initiation of CRT Xx Missing Xx Mean (SD) xx.x (xx.xx) Median xx.x (xx.xx) Median xx.x (xx.xx) Median xx.x (xx.xx) | Concurrent | |
| Missing Mean (SD) XX Median (SD) XX.X (min, max) (XX.XX, XX.XX) Number of cycles (Concurrent) n XX Missing XX Mean (SD) XX.X Median XX.X (min, max) (XX.XX, XX.XX) Tumor response assessment done on imaging (days) XX n XX Missing XX Mean (SD) XX.X (XX.XX) Median XX.X (min, max) (XX.XX, XX.XX) Performance status at time of initiation of CRT XX Missing XX Mean (SD) XX Mean (SD) XX Mean (SD) XX Median XX Median XXX Median XXX Median XXX | Number of cycles (Sequential) | |
| Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) Number of cycles (Concurrent) Xx n Xx Missing Xx Mean (SD) xx.x (xx.xx) Median (xx.xx, xx.xx) Median (xx.xx, xx.xx) In Xx Missing Xx Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) Performance status at time of initiation of CRT Xx n Xx Missing Xx Missing Xx Mean (SD) xx.x (xx.xx) Mean (SD) xx.x Mean (SD) xx.x (xx.xx) Median xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) | n | Xx |
| Median (min, max) xxxx Number of cycles (Concurrent) Xx n Xx Missing Xx Mean (SD) xxx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) Tumor response assessment done on imaging (days) Xx n Xx Missing Xx Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) Performance status at time of initiation of CRT Xx Missing Xx Mean (SD) xx.x (xx.xx) Median xx.x (xx.xx) xx.x Median xx.x (min, max) (xx.xx, xx.xx) | Missing | Xx |
| (min, max) (xx.xx, xx.xx) Number of cycles (Concurrent) Xx n Xx Missing Xx Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) Tumor response assessment done on imaging (days) Xx n Xx Missing Xx Median (SD) xx.x (xx.xx) (min, max) (xx.xx, xx.xx) Performance status at time of initiation of CRT Xx n Xx Missing Xx Mean (SD) xx.x (xx.xx) Median xx.x (min, max) xx.x | Mean (SD) | xx.x (xx.xx) |
| Number of cycles (Concurrent) Xx n Xx Missing Xx Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) Tumor response assessment done on imaging (days) Xx n Xx Missing Xx Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) Performance status at time of initiation of CRT Xx Missing Xx Mean (SD) xx.x Median xx.x Median xx.x (min, max) (xx.xx, xx.xx) | Median | xx.x |
| n Xx Missing Xx Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) Tumor response assessment done on imaging (days) Xx n Xx Missing Xx Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) Performance status at time of initiation of CRT Xx Missing Xx Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) | (min, max) | (xx.xx, xx.xx) |
| Missing Xx Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) Tumor response assessment done on imaging (days) Xx n Xx Missing Xx Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) Performance status at time of initiation of CRT Xx Missing Xx Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) | Number of cycles (Concurrent) | |
| Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) Tumor response assessment done on imaging (days) Xx n Xx Missing Xx Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) Performance status at time of initiation of CRT Xx Missing Xx Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) | n | Xx |
| Median (min, max) xx.x Tumor response assessment done on imaging (days) Xx N Xx Missing Xx Mean (SD) xx.x (xx.xx) Median xx.x (xx.xx) (min, max) (xx.xx, xx.xx) Performance status at time of initiation of CRT Xx Nissing Xx Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) | Missing | Xx |
| (min, max) (xx.xx, xx.xx) Tumor response assessment done on imaging (days) Xx n Xx Missing Xx Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) Performance status at time of initiation of CRT Xx n Xx Missing Xx Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) | Mean (SD) | xx.x (xx.xx) |
| Tumor response assessment done on imaging (days) Xx N Xx Missing Xx Median xx.x (min, max) (xx.xx, xx.xx) Performance status at time of initiation of CRT Xx N Xx Missing Xx Mean (SD) xx.x Median xx.x (min, max) (xx.xx, xx.xx) | Median | xx.x |
| n Xx Missing Xx Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) Performance status at time of initiation of CRT Xx n Xx Missing Xx Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) | (min, max) | (xx.xx, xx.xx) |
| Missing Xx Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) Performance status at time of initiation of CRT Xx n Xx Missing Xx Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) | Tumor response assessment done on imaging (days) | |
| Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) Performance status at time of initiation of CRT Xx n Xx Missing Xx Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) | n | Xx |
| Median xx.x (min, max) (xx.xx, xx.xx) Performance status at time of initiation of CRT Xx n Xx Missing Xx Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) | Missing | Xx |
| (min, max) (xx.xx, xx.xx) Performance status at time of initiation of CRT Xx n Xx Missing Xx Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) | • • | xx.x (xx.xx) |
| Performance status at time of initiation of CRT Xx n Xx Missing Xx Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) | Median | xx.x |
| n Xx Missing Xx Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) | (min, max) | (xx.xx, xx.xx) |
| Missing Xx Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) | Performance status at time of initiation of CRT | |
| Mean (SD) xx.x (xx.xx) Median xx.x (min, max) (xx.xx, xx.xx) | n | Xx |
| Median xx.x (min, max) (xx.xx, xx.xx) | Missing | Xx |
| (min, max) (xx.xx, xx.xx) | , , | xx.x (xx.xx) |
| | Median | xx.x |
| | | (xx.xx, xx.xx) |

- The Capital "N" in the column header represents the total number Enrolled Analysis Set.
- The small "n" represents the total number of patients in the row category.
- Percentages are based on total number of Enrolled Analysis Set.
- SD = Standard Deviation, min=minimum, max=maximum
- Source: Listing 16.1.9.1 and Listing 16.1.9.2



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|--------------------|
| Statistical Analysis Dlan | Version Number: | 3.1<br>25-Nov-2021 |
| Statistical Analysis Plan | Effective Date: | |

Table 14.1.8 Summary of WHO Performance Status (Safety Analysis Set)

| | N = xx |
|---|---|
| Visit 1 | |
| WHO Performance Grade | |
| 0 = Fully active, able to carry on all pre-disease performance without restriction | xx (xx.xx) |
| 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature | xx (xx.xx) |
| 2 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work | xx (xx.xx) |
| 3 = Capable of only limited self-care, confined to bed or chair more than 50% of waking hours | xx (xx.xx) |
| 4 = Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair | xx (xx.xx) |
| 5 = Dead | xx (xx.xx) |
| Visit x | |
| WHO Performance Grade | |
| 0 = Fully active, able to carry on all pre-disease performance without restriction | xx (xx.xx) |
| 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature | xx (xx.xx) |
| 2 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work | xx (xx.xx) |
| 3 = Capable of only limited self-care, confined to bed or chair more than 50% of waking hours | xx (xx.xx) |
| 4 = Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair | xx (xx.xx) |
| 5 = Dead | xx (xx.xx) |
| Patients performance grade changed, since last visit | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |

- The Capital "N" in the column header represents the total number of patients in Safety Analysis Set.
- The small "n" in summary statistic represents the total number of patients in the row category.
- Percentages are based on total number of patients in Safety Analysis Set.
- Programmer Note: Visit x- Visit 2 up to Visit 13.
- Source: Listing 16.1.10
- Table Name: xxxxx



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|---------|
| Statistical Analysis Plan | Version Number: | |
| Statistical Analysis Plan | Effective Date: | |

### Table 14.2.1.1 Adverse Events (Safety Analysis Set)

| | Durvalumab |
|---|---|
| | (N=xxx) |
| | n (%) E |
| Any Adverse Event | xx (xx.xx) xx |
| Any Serious Adverse Event | xx (xx.xx) xx |
| Any Treatment Emergent Adverse Event | xx (xx.xx) xx |
| Any Serious Treatment Emergent Adverse Event | xx (xx.xx) xx |
| Treatment Emergent Adverse Event related to IMP | xx (xx.xx) xx |
| Treatment Emergent Adverse Event leading to IMP discontinuation | xx (xx.xx) xx |
| Treatment Emergent Adverse Event leading to Death | xx (xx.xx) xx |

- The capital "N" in the column header represents the total number of patients in Safety Analysis Set.
- The small "n' in summary represents the number of patients in row category.
- TEAE are those adverse events which occurred after first dose of study medication.
- Note: Adverse events were coded using MedDRA version xx.x
- If a Patient has multiple occurrences of an AE, the Patient is presented only once in the respective patient count column (n)
  for the corresponding AE. Events are counted each time in the event (E)
- Source: Listing 16.3.1.1 and Listing 16.3.1.2



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|--------------------|
| Statistical Analysis Dlan | Version Number: | 3.1<br>25-Nov-2021 |
| Statistical Analysis Plan | Effective Date: | |

Table 14.2.1.2 Summary of Adverse Event (Safety Analysis Set)

| | Durvalumab<br>(N=xxx)<br>n (%) E |
|---|---|
| Any Adverse Event reported | xx (xx.xx) xx |
| Severity as per CTCAE grade | |
| Mild | xx (xx.xx) xx |
| Moderate | xx (xx.xx) xx |
| Severe | xx (xx.xx) xx |
| Life Threatening | xx (xx.xx) xx |
| Death | xx (xx.xx) xx |
| Action Taken to Study Drug | |
| No Change in IP | xx (xx.xx) xx |
| IP Temporarily Interrupted | xx (xx.xx) xx |
| IP Permanently Discontinued | xx (xx.xx) xx |
| Other | xx (xx.xx) xx |
| Treatment Given | |
| Yes | xx (xx.xx) xx |
| No | xx (xx.xx) xx |
| Relationship with Study Drug | . , |
| Related | xx (xx.xx) xx |
| Not Related | xx (xx.xx) xx |
| Outcome | |
| Resolved | xx (xx.xx) xx |
| Recovered/ Resolved with Sequelae | xx (xx.xx) xx |
| Recovering/ Resolving | xx (xx.xx) xx |
| Not Recovered/ Not Resolved | xx (xx.xx) xx |
| Fatal/ result in death | xx (xx.xx) xx |
| Unknown | xx (xx.xx) xx |
| Serious Adverse Event | |
| Yes | xx (xx.xx) xx |
| No | xx (xx.xx) xx |
| Seriousness Criteria | , |
| Death | xx (xx.xx) xx |
| Life-threatening | xx (xx.xx) xx |
| Inpatient hospitalization or prolongation of existing hospitalization | xx (xx.xx) xx |
| Document | |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Sandindinal Amelysis Plan | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

| Persistent or significant disability/ incapacity | xx (xx.xx) xx |
|--------------------------------------------------|---------------|
| Congenital anomaly/Birth Defect | xx (xx.xx) xx |
| Important medical events | xx (xx.xx) xx |
| Therapy Discontinued | |
| Yes | xx (xx.xx) xx |
| No | xx (xx.xx) xx |

- The Capital "N" in the column header represents the total number Safety Analysis Set.
- The small "n" represents the total number of patients in the row category.
- All Percentages rows are based on number of Safety Analysis Set.
- TEAE = treatment-emergent adverse event; E = number of TEAE
- All Percentages are based on the total number of Safety Analysis Set.
- Source: Listing 16.3.1.1 and Listing 16.3.1.2

Table 14.2.1.3 Summary of Treatment Emergent Adverse Events by System Organ Class and Preferred Term (Safety Analysis Set)

| | Durvalumab<br>(N=xxx) |
|----------------------|-----------------------|
| | n (%) E |
| Any TEAE | xx (xx.xx) xx |
| System Organ Class 1 | xx (xx.xx) xx |
| Preferred Term 1 | xx (xx.xx) xx |
| Preferred Term 2 | xx (xx.xx) xx |
| System Organ Class 2 | xx (xx.xx) xx |
| Preferred Term 1 | xx (xx.xx) xx |
| Preferred Term 2 | xx (xx.xx) xx |

- TEAE = treatment-emergent adverse event; N = number of Patients in the Safety Analysis Set; n = number of Patients with TEAE; E = number of TEAE
- All Percentages are based on the number of patients in Safety Analysis Set.
- System Organ Class and Preferred term are coded using MedDRA version xx.x
- System Organ classes and preferred term are sorted by descending frequency. Preferred terms are sorted by descending frequency within system organ class.
- Source: Listing 16.3.1.1 and Listing 16.3.1.2



| Document Title: | Document ID: | BP04-01 |
|----------------------------|-----------------|-------------|
| Statistical Applicate Plan | Version Number: | per: 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Table 14.2.1.4 Summary of Serious Treatment Emergent Adverse Events by System Organ Class and Preferred Term (Safety Analysis Set)

| | Durvalumab<br>(N=xxx) |
|----------------------|-----------------------|
| | n (%) E |
| Any Serious TEAE | xx (xx.xx) xx |
| System Organ Class 1 | xx (xx.xx) xx |
| Preferred Term 1 | xx (xx.xx) xx |
| Preferred Term 2 | xx (xx.xx) xx |
| System Organ Class 2 | xx (xx.xx) xx |
| Preferred Term 1 | xx (xx.xx) xx |
| Preferred Term 2 | xx (xx.xx) xx |

TEAE = treatment-emergent adverse event; N = number of Patients in the Safety Analysis Set; n = number of Patients with TEAE; E = number of TEAE

Source: Listing 16.3.1.1 and Listing 16.3.1.2

<sup>-</sup> All Percentages are based on the total number of patients in Safety Analysis Set.

<sup>-</sup> System Organ Class and Preferred term are coded using MedDRA version xx.x

System Organ classes and preferred term are sorted by descending frequency. Preferred terms are sorted by descending frequency within system organ class.



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.2.1.5 Summary of Treatment Emergent Adverse Events leading to permanent discontinuation by System Organ Class and Preferred Term (Safety Analysis Set)

| | Durvalumab<br>(N=xxx) |
|-----------------------------------------------|-----------------------|
| | n (%) E |
| Any TEAE leading to permanent discontinuation | xx (xx.xx) xx |
| System Organ Class 1 | xx (xx.xx) xx |
| Preferred Term 1 | xx (xx.xx) xx |
| Preferred Term 2 | xx (xx.xx) xx |
| System Organ Class 2 | xx (xx.xx) xx |
| Preferred Term 1 | xx (xx.xx) xx |
| Preferred Term 2 | xx (xx.xx) xx |

TEAE = treatment-emergent adverse event; N = number of Patients in the Safety Analysis Set; n = number of Patients with TEAE; E = number of TEAE

- All Percentages are based on the total number of patients in Safety Analysis Set.
- System Organ Class and Preferred term are coded using MedDRA version xx.x
- System Organ classes and preferred term are sorted by descending frequency. Preferred terms are sorted by descending frequency within system organ class.
- Source: Listing 16.3.1.1 and Listing 16.3.1.2



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.2.1.6 Summary of Treatment Emergent Adverse Events leading to Death by System Organ Class and Preferred Term (Safety Analysis Set)

| | Durvalumab<br>(N=xxx) |
|---------------------------|-----------------------|
| | n (%) E |
| Any TEAE leading to death | xx (xx.xx) xx |
| System Organ Class 1 | xx (xx.xx) xx |
| Preferred Term 1 | xx (xx.xx) xx |
| Preferred Term 2 | хх (хх.хх) хх |
| System Organ Class 2 | xx (xx.xx) xx |
| Preferred Term 1 | xx (xx.xx) xx |
| Preferred Term 2 | xx (xx.xx) xx |

TEAE = treatment-emergent adverse event; N = number of Patients in the Safety Analysis Set; n = number of Patients with TEAE; E = number of TEAE

- All Percentages are based on the total number of patients in Safety Analysis Set.
- System Organ Class and Preferred term are coded using MedDRA version xx.x
- System Organ classes and preferred term are sorted by descending frequency. Preferred terms are sorted by descending frequency within system organ class.
- Source: Listing 16.3.1.1 and Listing 16.3.1.2



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.2.1.7 Summary of Treatment Emergent Adverse Event by System Organ Class, Preferred Term and Severity (Safety Analysis Set)

| | Durvalumab<br>(N=xxx) | | | | |
|---|---|---|---|---|---|
| | Mild | Mild Moderate Severe Life Threatening | | | |
| | n (%) E | n (%) E | n (%) E | n (%) E | n (%) E |
| Any TEAE | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx |
| System Organ Class 1 | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx |
| Preferred Term 1 | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx |
| Preferred Term 2 | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx |
| System Organ Class 2 | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx |
| Preferred Term 1 | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx |
| Preferred Term 2 | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx |

TEAE = treatment-emergent adverse event; N = number of Patients in the Safety Analysis Set; n = number of Patients with TEAE; E = number of TEAE

<sup>-</sup> All Percentages are based on the total number of patients in Safety Analysis Set.

System Organ Class and Preferred term are coded using MedDRA version xx.x

System Organ classes and preferred term are sorted by descending frequency. Preferred terms are sorted by descending frequency within system organ class.

Source: Listing 16.3.1.1 and Listing 16.3.1.2



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.2.1.8 Summary of Treatment Emergent Adverse Event by System Organ Class and Preferred Term (Safety Analysis Set)

| | Durvalumab |
|----------------------|---------------|
| | (N=xxx) |
| | Related |
| | n (%) E |
| Any Related TEAE | xx (xx.xx) xx |
| System Organ Class 1 | xx (xx.xx) xx |
| Preferred Term 1 | xx (xx.xx) xx |
| Preferred Term 2 | xx (xx.xx) xx |
| System Organ Class 2 | xx (xx.xx) xx |
| Preferred Term 1 | xx (xx.xx) xx |
| Preferred Term 2 | xx (xx.xx) xx |

TEAE = treatment-emergent adverse event; N = number of Patients in the Safety Analysis Set; n = number of Patients with TEAE; E = number of TEAE

- All Percentages are based on the total number of patients in Safety Analysis Set.
- System Organ Class and Preferred term are coded using MedDRA version xx.x
- System Organ classes and preferred term are sorted by descending frequency. Preferred terms are sorted by descending frequency within system organ class.
- Source: Listing 16.3.1.1 and Listing 16.3.1.2

Table 14.2.1.9 Summary of Serious Treatment Emergent Adverse Event by System Organ Class and Preferred Term (Safety Analysis Set)

| | Durvalumab |
|--------------------------|---------------|
| _ | (N=xxx) |
| | Related |
| | n (%) E |
| Any Related Serious TEAE | xx (xx.xx) xx |
| System Organ Class 1 | xx (xx.xx) xx |
| Preferred Term 1 | xx (xx.xx) xx |
| Preferred Term 2 | xx (xx.xx) xx |
| System Organ Class 2 | xx (xx.xx) xx |
| Preferred Term 1 | xx (xx.xx) xx |
| Preferred Term 2 | xx (xx.xx) xx |

TEAE = treatment-emergent adverse event; N = number of Patients in the Safety Analysis Set; n = number of Patients with TEAE; E = number of TEAE

System Organ classes and preferred term are sorted by descending frequency. Preferred terms are sorted by descending frequency within system organ class.

| Document |
|---------------------------------------|
|---------------------------------------|

All Percentages are based on the total number of patients in Safety Analysis Set.

System Organ Class and Preferred term are coded using MedDRA version xx.x



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Source: Listing 16.3.1.1 and Listing 16.3.1.2

Table 14.2.1.10 Summary of Treatment Emergent Adverse Event by System Organ Class, Preferred Term and Relationship with Study Drug (Safety Analysis Set)

| | Durvalumab | | | | | |
|---|---|---|---|---|---|---|
| | (N=xxx) | | | | | |
| | | Resolve with Resolving Not Resolved Result in | | | | |
| | Resolved | Sequelae | | | Death | |
| | n (%) E | n (%) E | n (%) E | n (%) E | n (%) E | n (%) E |
| Any TEAE | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx |
| System Organ Class 1 | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx |
| Preferred Term 1 | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx |
| Preferred Term 2 | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx |
| System Organ Class 2 | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx |
| Preferred Term 1 | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx |
| Preferred Term 2 | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx | xx (xx.xx) xx |

- TEAE = treatment-emergent adverse event; N = number of Patients in the Safety Analysis Set; n = number of Patients with TEAE; E = number of TEAE
- All Percentages are based on the total number of patients in Safety Analysis Set.
- System Organ Class and Preferred term are coded using MedDRA version xx.x
- System Organ classes and preferred term are sorted by descending frequency. Preferred terms are sorted by descending frequency within system organ class.
- Source: Listing 16.3.1.1 and Listing 16.3.1.2


| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Shakishing Angloria Plan | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Table 14.3.1 Summary of Physical Examination (Safety Analysis Set)

| | Durvalumab |
|---------------------------------------|-----------------|
| | N = xx<br>n (%) |
| Visit x | 11 (70) |
| Patients Examination Done | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| Missing | xx (xx.xx) |
| General Appearance | ^^ (^^.^^) |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | ^^ (^^.^^) |
| NCS | xx (xx.xx) |
| CS | xx (xx.xx) |
| | ** (**.**) |
| Respiratory Normal | w /w w/ |
| Abnormal | xx (xx.xx) |
| If Abnormal | xx (xx.xx) |
| NCS | and the second |
| | xx (xx.xx) |
| CS<br>Continuous I o | xx (xx.xx) |
| Cardiovascular | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | , |
| NCS | xx (xx.xx) |
| CS | xx (xx.xx) |
| Abdomen | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | |
| NCS | xx (xx.xx) |
| CS | xx (xx.xx) |
| Skin | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | |
| NCS | xx (xx.xx) |
| CS | xx (xx.xx) |
| HEENT | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | |
| NCS | xx (xx.xx) |
| CS | xx (xx.xx) |
| Neck | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| Document | |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

| If Almontol | |
|---|---|
| If Abnormal | () |
| NCS | xx (xx.xx) |
| CS | xx (xx.xx) |
| Lymph Node | , , |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | |
| NCS | xx (xx.xx) |
| CS | xx (xx.xx) |
| Thyroid | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | |
| NCS | xx (xx.xx) |
| CS | xx (xx.xx) |
| Musculo-skeletal | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | |
| NCS | xx (xx.xx) |
| CS | xx (xx.xx) |
| Genital/Rectal | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | |
| NCS | xx (xx.xx) |
| CS | xx (xx.xx) |
| Neurological | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | |
| NCS | xx (xx.xx) |
| CS | xx (xx.xx) |
| Others | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | |
| NCS | xx (xx.xx) |
| CS | xx (xx.xx) |
| The Control WAII in the column hander common to the text of control of Coffee Analysis Coffee | |

- The Capital "N" in the column header represents the total number Safety Analysis Set.
- The small "n" represents the total number of patients in the row category.
- All Percentages rows are based on number of Safety Analysis Set.
- Programmer Note: Visit x Visit 1 up to Visit 12.
- Source: Listing 16.3.2



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.3.2 Summary of Vital Sign (Safety Analysis Set)

| | N = xx |
|---------------------------------|----------------|
| Visit x | |
| Examination Done, n (%) | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| Missing | xx (xx.xx) |
| Systolic Blood Pressure (mmHg) | |
| n | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |
| Diastolic Blood Pressure (mmHg) | |
| n | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |
| Pulse Rate (beats/min) | |
| n | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |
| Respiratory Rate (breaths/min) | |
| n | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |
| Temperature (°F) | |
| n | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |
| Oxygen Saturation (%) | |
| n | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |
| Weight (Kg) | |
| n | Xx |
| Missing | Xx |


** Document** 



| Document Title: | Document ID: | BP04-01 |
|-----------------------------|-----------------|-------------|
| Statistical Applicate Plans | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

 Mean (SD)
 xx.x (xx.xx)

 Median
 xx.x

 (min, max)
 (xx.xx, xx.xx)

- The Capital "N" in the column header represents the total number Safety Analysis Set.
- The small "n" represents the total number of patients in the row category.
- Percentages in the "Examination Done" rows are based on number of Safety Analysis Set.
- SD = Standard Deviation, min=minimum, max=maximum
- Programmer Note: Visit x Visit 2 up to Visit 12.
- Source: Listing 16.3.3



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.3.3 Summary of 12-Lead Electrocardiogram (Safety Analysis Set)

| | N = xx |
|------------------------|----------------|
| Visit x | |
| Assessment Done, n (%) | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| Missing | xx (xx.xx) |
| Heart rate (beats/min) | |
| n | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |
| QRS (ms) | |
| n | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | XX.X |
| (min, max) | (xx.xx, xx.xx) |
| PR (ms) | |
| n | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |
| RR (ms) | |
| n | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |
| QT (ms) | |
| n | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |
| QTcF (ms) | |
| n | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |

- The Capital "N" in the column header represents the total number Safety Analysis Set.
- The small "n" represents the total number of patients in the row category.
- Percentages in the "Assessment Done" rows are based on number of Safety Analysis Set.
- SD = Standard Deviation, min=minimum, max=maximum



| | Document Title: | Document ID: | BP04-01 |
|---|---|---|---|
| Chatletteel Academic Plans | Version Number: | 3.1 | |
| | Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Programmer Note: Visit x – Visit 2, Visit 6 and Visit 10.

Source: Listing 16.3.4



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Shakishing Angloria Plan | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Table 14.3.4.1 Summary of Haematology (Safety Analysis Set)

| | N = xx |
|---------------------------------------|---------------|
| | n (%) |
| Visit x | |
| Sample Collected | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| Missing | xx (xx.xx) |
| Haematocrit | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |
| Haemoglobin | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| lf Abnormal | |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |
| Basophils | • |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| f Abnormal | . , |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |
| Eosinophils | , , |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | , |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |
| Monocytes | , |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| f Abnormal | |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |
| Absolute Neutrophil Count | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |
| Platelet count | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| f Abnormal | 00 (00:00) |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |
| Total Lymphocyte count | 00 (00:00) |
| Document | |



| Document Title: | Document ID: | BP04-01 |
|-----------------|--------------|---------|
| Effective Date: | 25-Nov-2021 | |

| Normal | xx (xx.xx) |
|-------------------------------|------------|
| Abnormal | xx (xx.xx) |
| If Abnormal | |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |
| Differential Lymphocyte count | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |

- The Capital "N" in the column header represents the total number Safety Analysis Set.
- The small "n" represents the total number of patients in the row category.
- All Percentages rows are based on number of Safety Analysis Set.
- NCS=Abnormal Not Clinically Significant and CS= Abnormal Clinically Significant
- Programmer Note: Visit x Visit 2 up to Visit 12.
- Source: Listing 16.3.5



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.3.4.2 Summary of Serum Chemistry (Safety Analysis Set)

| | N = xx |
|---------------------------------------|---------------|
| | n (%) |
| Visit x | |
| Sample Collected | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| Missing | xx (xx.xx) |
| Albumin | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |
| Glucose | , , |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |
| Alkaline phosphatase | on funion) |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | an (anian) |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |
| Lactate dehydrogenase | ^^ (^^.^^) |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| f Abnormal | ** (**.**) |
| CS | yy /yy yyl |
| NCS | xx (xx.xx) |
| Alanine aminotransferase | xx (xx.xx) |
| Normal | |
| Abnormal | xx (xx.xx) |
| | xx (xx.xx) |
| f Abnormal | |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |
| Lipase | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| lf Abnormal | |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |
| Aspartate amin-otransferase | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| f Abnormal | |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |
| Magnesium | |
| Document | Dogo 45 of 77 |
| Document | |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

| Document | |
|---|---|
| Desument | Dago 46 -677 |
| CS | xx (xx.xx) |
| If Abnormal | |
| Abnormal | xx (xx.xx) |
| Normal | xx (xx.xx) |
| Total protein | |
| NCS | xx (xx.xx) |
| CS | xx (xx.xx) |
| If Abnormal | |
| Abnormal | xx (xx.xx) |
| Normal | xx (xx.xx) |
| Chloride | |
| NCS | xx (xx.xx) |
| CS | xx (xx.xx) |
| If Abnormal | , , |
| Abnormal | xx (xx.xx) |
| Normal | xx (xx.xx) |
| Total bilirubin | , |
| NCS | xx (xx.xx) |
| CS | xx (xx.xx) |
| If Abnormal | an (anian) |
| Abnormal | xx (xx.xx) |
| Normal | xx (xx.xx) |
| NCS<br>Calcium | xx (xx.xx) |
| CS<br>NCS | xx (xx.xx) |
| If Abnormal | |
| Abnormal | xx (xx.xx) |
| Normal | xx (xx.xx) |
| Sodium | |
| NCS | xx (xx.xx) |
| CS | xx (xx.xx) |
| If Abnormal | |
| Abnormal | xx (xx.xx) |
| Normal | xx (xx.xx) |
| Bicarbonate | |
| NCS | xx (xx.xx) |
| CS | xx (xx.xx) |
| If Abnormal | |
| Abnormal | xx (xx.xx) |
| Normal | xx (xx.xx) |
| Potassium | |
| NCS | xx (xx.xx) |
| CS | xx (xx.xx) |
| If Abnormal | |
| Abnormal | xx (xx.xx) |
| Normal | xx (xx.xx) |
| Amylase | · |
| NCS | xx (xx.xx) |
| CS | xx (xx.xx) |
| If Abnormal | ( |
| Abnormal | xx (xx.xx) |
| Normal | xx (xx.xx) |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

| NCS | xx (xx.xx) |
|-----------------------------|-----------------------------------------|
| Creatinine Clearance | na (man) |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | in (initial) |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |
| Urea / Blood Urea/ Nitrogen | , |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | , |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |
| Gamma glutamyl transferase | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |
| Uric acid | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |

- The Capital "N" in the column header represents the total number Safety Analysis Set.
- The small "n" represents the total number of patients in the row category.
- All Percentages rows are based on number of Safety Analysis Set.
- NCS=Abnormal Not Clinically Significant and CS= Abnormal Clinically Significant
- Programmer Note: Visit x Visit 2 up to Visit 12.
- Source: Listing 16.3.6



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.3.4.3 Summary of Urine Routine and Microscopy (Safety Analysis Set)

| | N = xx |
|---------------------------------------|--------------------------|
| | n (%) |
| Visit x | |
| Sample Collected | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| Missing | xx (xx.xx) |
| Specific gravity | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |
| pH | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| lf Abnormal | |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |
| Glucose | , |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| lf Abnormal | , |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |
| Ketones | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| f Abnormal | an (aman) |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |
| Bilirubin | an (anian) |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| f Abnormal | ~~ (~~~~) |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |
| Urobilinogen | ** (**.**) |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx)<br>xx (xx.xx) |
| If Abnormal | ** (**.**) |
| CS CS | vu lvu vul |
| NCS | xx (xx.xx) |
| RBC | xx (xx.xx) |
| Normal | www.free.com |
| Abnormal | xx (xx.xx) |
| | xx (xx.xx) |
| If Abnormal | t |
| CS<br>NCS | xx (xx.xx) |
| NCS | xx (xx.xx) |
| Dysmorphic Red Blood Cells | |
| Document | |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

| Normal | xx (xx.xx) |
|---|---|
| Abnormal | xx (xx.xx) |
| If Abnormal | |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |
| Pus Cells | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |
| Crystals | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | . , |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |
| Casts | , |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | , , |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |
| Epithelial Cells | , |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |
| Protein | , |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |
| The Control Hall is also asked to be added to the standard to the Control Cont | |

- The Capital "N" in the column header represents the total number Safety Analysis Set.
- The small "n" represents the total number of patients in the row category.
- All Percentages rows are based on number of Safety Analysis Set.
- NCS=Abnormal Not Clinically Significant and CS= Abnormal Clinically Significant
- Programmer Note: Visit x Visit 2 up to Visit 12.
- Source: Listing 16.3.7



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.3.4.4 Summary of Thyroid function test (Safety Analysis Set)

| | N = xx |
|---------------------|------------|
| | n (%) |
| Visit x | |
| Sample Collected | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| Missing | xx (xx.xx) |
| TSH | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |
| Tri iodothyronine | |
| Not applicable | xx (xx.xx) |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |
| Tetra iodothyronine | |
| Not Applicable | xx (xx.xx) |
| Normal | xx (xx.xx) |
| Abnormal | |
| If Abnormal | |
| CS | xx (xx.xx) |
| NCS | xx (xx.xx) |

- The Capital "N" in the column header represents the total number Safety Analysis Set.
- The small "n" represents the total number of patients in the row category.
- All Percentages rows are based on number of Safety Analysis Set.
- NCS=Abnormal Not Clinically Significant and CS= Abnormal Clinically Significant
- Programmer Note: Visit x Visit 2, Visit 6, Visit 10 and Visit 12.
- Source: Listing 16.3.8

Table 14.3.5 Summary of Urine Pregnancy Test (Safety Analysis Set - Female)

| Visit | | Durvalumab<br>N* = xx |
|---|---|---|
| | • | n (%) |
| Visit 1 | Numbe of patients' urine pregnancy test | |
| | performed | |
| | Yes | xx (xx.xx) |
| | No | xx (xx.xx) |
| | NA | xx (xx.xx) |
| | Result | |
| Proprietary an | d Confidential Document | |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Blan | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

| | Positive | xx (xx.xx) |
|---------|---------------------------------------------------|------------|
| | Negative | xx (xx.xx) |
| Visit 2 | Numbe of patients' urine pregnancy test performed | |
| | Yes | xx (xx.xx) |
| | No | xx (xx.xx) |
| | NA | xx (xx.xx) |
| | Result | |
| | Positive | xx (xx.xx) |
| | Negative | xx (xx.xx) |

.....

- The Capital "N" in the column header represents the total number Enrolled Analysis Set.
- The small "n" represents the total number of patients in the row category.
- Percentages in the "Urine pregnancy test performed" rows are based on number of Enrolled Analysis Set.
- Percentages in the "Result" rows are based on number of patient urine pregnancy test performed.
- Source: Listing 16.1.7



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# Listings

Listing 16.1.1.1. Listing of Patient Informed Consent Details

| Unique Patient | Informed | Date and Time for | Subject | Audio-visual consent |
|---|---|---|---|---|
| ID | Consent taken | Informed Consent | vulnerable | taken |
| Xxxxxx | Yes/No | DD-MMM-YYYY/HH:MM | Yes/No | Yes/No |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Listing 16.1.1.2 Listing of Patient Eligibility Criteria and Analysis Population Set

| Unique Patient<br>ID | Patients Subject<br>meet all Enrolled<br>Eligibility into the<br>Criteria Study | | meet all Enrolled Eligibility into the | | Safety Analysis Set |
|---|---|---|---|---|---|
| Xxxxxx | Yes/No | Yes/No | Yes/No | Yes/No | |
| Xxxxxx | Yes/No | Yes/No | Yes/No | Yes/No | |
| Xxxxxx | Yes/No | Yes/No | Yes/No | Yes/No | |
| Xxxxxx | Yes/No | Yes/No | Yes/No | Yes/No | |
| Xxxxxx | Yes/No | Yes/No | Yes/No | Yes/No | |

#### Listing 16.1.1.3 Listing of Patient Study Completion / Discontinuation

| Unique | Patient completed the | Date of study | Primary reason of |
|---|---|---|---|
| Patient ID | study | completion/discontinuation | Discontinuation |
| XXXXXX | Yes/No | DD-MMM-YYYY | XXXX |
| XXXXXX | Yes/No | DD-MMM-YYYY | XXXX |
| XXXXXX | Yes/No | DD-MMM-YYYY | XXXX |
| XXXXXX | Yes/No | DD-MMM-YYYY | Other: xxxxx |
| XXXXXX | Yes/No | DD-MMM-YYYY | xxxx |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Listing 16.1.1.4 Listing of Patient Protocol Deviation

| Unique | Patient undergone any | Sr. | | Date of study | | Deviation | Action |
|---|---|---|---|---|---|---|---|
| Patient ID | <b>Protocol Deviation</b> | no | Deviation | Deviation | Description | Code | taken |
| XXXXXX | Yes/No | Xx | XXXX | DD-MMM-YYYY | XXXX | Xx | Xx |
| XXXXX | Yes/No | Xx | XXXX | DD-MMM-YYYY | XXXX | Xx | Xx |
| XXXXXX | Yes/No | Xx | XXXX | DD-MMM-YYYY | XXXX | Xx | Xx |
| XXXXXX | Yes/No | Xx | XXXX | DD-MMM-YYYY | XXXX | Xx | Xx |
| xxxxx | Yes/No | Xx | XXXX | DD-MMM-YYYY | XXXX | Xx | Xx |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Blan | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

#### Listing 16.1.2 Listing of Patient Demographics Data

| Unique Patient<br>ID | Age / Gender | Date of Birth | Weight (kg) | Height (cm) | Race | If Other |
|---|---|---|---|---|---|---|
| XXXXXX | xx/xxx | DD-MMM-YYYY | XXX | XXX | Indian/Other | XXXX |
| XXXXXX | xx/xxx | DD-MMM-YYYY | XXX | xxx | Indian/Other | XXXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Listing 16.1.3 Listing of Patient Medical / Surgical History

| Unique | MH. | Medical/Surgical | Type of | System Organ | Preferred Term | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Patient ID | No | history | Condition | Class | | Start date | Stop date | Treatment | Ongoing |
| | | | | | | | | Required | |
| XXXXXX | XXX | XXX | XXX | XXX | XXX | DD-MMM- | DD-MMM- | Yes/No | XXX |
| | | | | | | YYYY | YYYY | | |
| XXXXXX | xxx | xxx | xxx | xxx | xxx | DD-MMM- | DD-MMM- | Yes/No | XXX |
| | | | | | | YYYY | YYYY | | |
| XXXXXX | XXX | XXX | xxx | XXX | XXX | DD-MMM- | DD-MMM- | Yes/No | XXX |
| | | | | | | YYYY | YYYY | | |
| XXXXXX | XXX | XXX | XXX | XXX | XXX | DD-MMM- | DD-MMM- | Yes/No | XXX |
| | | | | | | YYYY | YYYY | | |
| XXXXXX | xxx | XXX | xxx | xxx | XXX | DD-MMM- | DD-MMM- | Yes/No | xxx |
| | | | | | | YYYY | YYYY | | |

Patients with at least one medical/ Surgical History have been listed.



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Applyais Plan | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

#### Listing 16.1.4.1 Listing of Patient IP Administration I

| Unique | | | Days of completion of CRT durvalumab | Total Dose | Stop Time of Infusion |
|---|---|---|---|---|---|
| Patient ID | Visit | Date and Time of Infusion of IP | Started | (mg/mL) | of IP |
| XXXXXXX | XXX | DD-MMM-YYYY/HH:MM | xxx | XXX | XXX |
| XXXXXX | XXX | DD-MMM-YYYY/HH:MM | xxx | XXX | XXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Applyais Plan | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

# Listing 16.1.4.2 Listing of Patient IP Administration II

| Unique | | Dose interrupted during | If | Interruption time | Dose | If | If Yes, Provide the restart |
|---|---|---|---|---|---|---|---|
| Patient ID | Visit | infusion | yes | | Restated | No | time |
| xxxxxx | XXX | Yes/No | XXX | DD-MMM-YYYY | Yes/No | xxx | xxx |
| xxxxx | XXX | Yes/No | XXX | DD-MMM-YYYY | Yes/No | XXX | xxx |
| xxxxx | XXX | Yes/No | XXX | DD-MMM-YYYY | Yes/No | XXX | xxx |
| XXXXXX | XXX | Yes/No | XXX | DD-MMM-YYYY | Yes/No | XXX | XXX |
| xxxxxx | XXX | Yes/No | XXX | DD-MMM-YYYY | Yes/No | XXX | XXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# Listing 16.1.4.3. Listing of Patient Study Drug Administration Accountability

| Unique | Dose reduced in | If | If Yes, Visit | Dose | If | No. of IV Dose has to administered | No. of IV Dose has to administered | Unused IP | Compliance |
|---|---|---|---|---|---|---|---|---|---|
| Patient | any of the visit | yes | number | Competed | No | during treatment period | in the treatment period | returned | (%) |
| ID | | | | | | | | | |
| XXXXXX | Yes/No | XXX | XXX | Yes/No | XXX | xxx | xxx | Yes/No | XXX |
| XXXXXX | Yes/No | XXX | XXX | Yes/No | XXX | xxx | XXX | Yes/No | XXX |
| XXXXXXX | Yes/No | XXX | XXX | Yes/No | XXX | xxx | xxx | Yes/No | XXX |
| XXXXXXX | Yes/No | XXX | XXX | Yes/No | XXX | xxx | xxx | Yes/No | XXX |
| XXXXXXX | Yes/No | XXX | XXX | Yes/No | XXX | xxx | xxx | Yes/No | XXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Chabinhinal Analysis Blan | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Listing 16.1.5 Listing of Patient Disease characteristics Assessment

| Unique Patient<br>ID | Visit | Disease Staging | Disease progressed since last visit |
|---|---|---|---|
| xxxxxx | xxx | XXX | Yes/No |
| XXXXXX | XXX | XXX | Yes/No |
| XXXXXX | XXX | XXX | Yes/No |
| XXXXXX | XXX | XXX | Yes/No |
| xxxxx | xxx | XXX | Yes/No |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Listing 16.1.6.1 Listing of Patient Alcohol consumption and drug abuse

| Unique Patient | Patient have any significant history | If Yes, | | If Yes, Drug | |
|---|---|---|---|---|---|
| ID | of alcoholism or drug abuse | Alcohol | Quit date | abuse | Quit date |
| xxxxxx | Yes/No | XXX | DD-MMM-YYYY | XXX | DD-MMM-YYYY |
| XXXXXXX | Yes/No | XXX | DD-MMM-YYYY | XXX | DD-MMM-YYYY |
| XXXXXXX | Yes/No | XXX | DD-MMM-YYYY | XXX | DD-MMM-YYYY |
| XXXXXX | Yes/No | XXX | DD-MMM-YYYY | XXX | DD-MMM-YYYY |
| XXXXXX | Yes/No | XXX | DD-MMM-YYYY | xxx | DD-MMM-YYYY |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# Listing 16.1.6.2 Listing of Patient History of Tobacco

| Unique Patient ID | Smoking History |
|-------------------|-----------------|
| xxxxxx | xxx |
| xxxxxx | XXX |
| XXXXXX | XXX |
| XXXXXX | XXX |
| XXXXXX | XXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Listing 16.1.7 Listing of Patient Urine Pregnancy Test

| Unique | Visit | Urine pregnancy test | Date and Time of | Result |
|---|---|---|---|---|
| Patient ID | | performed | Assessment | |
| XXXXXX | Visit 1 | Yes/No/NA | DD-MMM-YYYY | Positive/Negative |
| | Visit 2 | Yes/No/NA | DD-MMM-YYYY | Positive/Negative |
| | | Yes/No/NA | DD-MMM-YYYY | Positive/Negative |
| XXXXXX | Visit 1 | Yes/No/NA | DD-MMM-YYYY | Positive/Negative |
| | | Yes/No/NA | DD-MMM-YYYY | Positive/Negative |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Listing 16.1.8 Listing of Patient Prior/Concomitant Medications

| Unique<br>Patient<br>ID | Medication<br>Name<br>(Generic) | ATC<br>Drug<br>Class | Standard<br>Name | Start Date<br>-End<br>Date/Ongoing | Indication | Dosage<br>Form | Dose<br>(unit) | Route | Frequency |
|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXXX | XXXX | XXXX | DDMMYYYY- | XXX | xx | xx (xx) | XXXX | XX |
| XXXXXX | Xxx xxx | XXXXX | xxxxx | DDMMYYYY<br>DDMMYYYY- | xxx | xxxx | xx (xx) | xxxx | хххх |
| xxxxx | Xxx xxxx | XXXX | XXXX | Ongoing<br>DDMMYYYY-<br>DDMMYYYY | xx | xxx | xx (xx) | xxxx | xxx |
| xxxxx | Xxxxx xxxxx | xxxx | xxxxx | DDMMYYYY-<br>DDMMYYYY | xx | xxx | xx (xx) | xxxx | xx |
| xxxxx | XXXXXXXXXXX | XXXX | XXXX | DDMMYYYY-<br>Ongoing | xx | xxx | xx (xx) | xxxx | xxx |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

#### Listing 16.1.9.1 Listing of Patient Radiation Treatment

| Unique | Clinical Stage of | Pathological Staging of | Pathological Staging | Histology of | Technique of | Dose of | Chemotherapy | If | No. Of |
|---|---|---|---|---|---|---|---|---|---|
| Patient ID | NSCLC | NSCLC done | of NSCLC | Tumor | Radiation | Radiation | given | Yes | Cycles |
| xxxxx | xxx | Yes/No | XXX | XXX | xxx | XXX | Yes/No | XXX | xxx |
| xxxxx | xxx | Yes/No | XXX | XXX | xxx | xxx | Yes/No | XXX | xxx |
| XXXXX | XXX | Yes/No | XXX | XXX | XXX | XXX | Yes/No | XXX | xxx |
| XXXXX | xxx | Yes/No | XXX | XXX | xxx | XXX | Yes/No | XXX | xxx |
| xxxxx | xxx | Yes/No | XXX | Xxx | Xxx | Xxx | Yes/No | Xxx | Xxx |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# Listing 16.1.9.2 Listing of Patient Radiation Treatment

| Unique Patient | Type of | Chemo | No. of | Days of CRT | Performance status at time of |
|---|---|---|---|---|---|
| ID | Chemotherapy | regime | Cycles | | initiation of CRT |
| xxxxxx | xxx | XXX | XXX | xxx | xxx |
| XXXXXX | xxx | XXX | XXX | xxx | XXX |
| XXXXXX | XXX | XXX | XXX | xxx | XXX |
| XXXXXX | XXX | XXX | XXX | xxx | XXX |
| XXXXXX | XXX | XXX | XXX | XXX | XXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# Listing 16.1.10 Listing of Patient WHO Performance status

| Unique Patient<br>ID | Visit | Туре | WHO Performance Grade | If there any changes in performance grade since last visit |
|---|---|---|---|---|
| xxxxxx | xxx | XXX | xxx | Yes/No |
| XXXXXX | XXX | XXX | xxx | Yes/No |
| XXXXXX | XXX | XXX | xxx | Yes/No |
| XXXXXX | XXX | XXX | xxx | Yes/No |
| XXXXXX | XXX | XXX | xxx | Yes/No |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

#### Listing 16.3.1.1 Listing of Patient Adverse Event

| Unique Patient | Visit | Patient have any Adverse | Patient have any Adverse |
|---|---|---|---|
| ID | | Event since screening visit | <b>Event since last visit</b> |
| xxxxxx | XXX | Yes/No | Yes/No |
| xxxxxx | xxx | Yes/No | Yes/No |
| xxxxxx | XXX | Yes/No | Yes/No |
| xxxxxx | XXX | Yes/No | Yes/No |
| XXXXXX | XXX | Yes/No | Yes/No |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

#### Listing 16.3.1.2 Listing of Patient Adverse Event

| Unique | Adverse | AE No. | Adverse Event | System organ | Preferred | Start Date and time | Stop Date and time | Severity as per | Action taken |
|---|---|---|---|---|---|---|---|---|---|
| Patient | Event | | Term | class | Term | | | CTCAE grade | |
| ID | | | | | | | | | |
| xxxxxx | Yes/No | XXX | XXX | xxx | XXX | DD-MMM-YYYY/HH:MM | DD-MMM-YYYY/HH:MM | xx | xxx |
| XXXXXX | Yes/No | XXX | XXX | xxx | XXX | DD-MMM-YYYY/HH:MM | DD-MMM-YYYY/HH:MM | Xx | xxx |
| xxxxxx | Yes/No | XXX | XXX | xxx | XXX | DD-MMM-YYYY/HH:MM | DD-MMM-YYYY/HH:MM | XX | xxx |
| XXXXXX | Yes/No | XXX | XXX | xxx | XXX | DD-MMM-YYYY/HH:MM | DD-MMM-YYYY/HH:MM | XX | xxx |
| XXXXXX | Yes/No | XXX | xxx | xxx | xxx | DD-MMM-YYYY/HH:MM | DD-MMM-YYYY/HH:MM | xx | xxx |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Listing 16.3.1.3 Listing of Patient Adverse Event

| Unique | Adverse | AE No. | Adverse Event | Treatment | Relationship | Outcome | Serious AE | Therapy |
|---|---|---|---|---|---|---|---|---|
| Patient | Event | | Term | given | with study Drug | | | Discontinued |
| ID | | | | | | | | |
| XXXXXXX | Yes/No | XXX | XXX | Yes/No | XXX | XXX | Yes/No | Yes/No |
| XXXXXXX | Yes/No | XXX | XXX | Yes/No | XXX | XXX | Yes/No | Yes/No |
| XXXXXXX | Yes/No | XXX | XXX | Yes/No | XXX | XXX | Yes/No | Yes/No |
| XXXXXX | Yes/No | XXX | XXX | Yes/No | XXX | XXX | Yes/No | Yes/No |
| XXXXXX | Yes/No | XXX | xxx | Yes/No | XXX | XXX | Yes/No | Yes/No |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Listing 16.3.2 Listing of Patient Physical Examination

| Unique<br>Patient<br>ID | Visit | Examination<br>done | Date and Time of<br>Assessment | Physical<br>Examination | Result | If<br>Abnormal |
|---|---|---|---|---|---|---|
| XXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | XXX | Normal/Abnormal | CS/NCS |
| XXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | XXX | Normal/Abnormal | CS/NCS |
| XXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | XXX | Normal/Abnormal | CS/NCS |
| XXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | xxx | Normal/Abnormal | CS/NCS |
| XXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | xxx | Normal/Abnormal | CS/NCS |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Listing 16.3.3 Listing of Patient Vital Signs

| Unique Patient | Visit | Examination Done | Date and Time of Assessment | Parameter | Result | Assessment Result | If Abnormal |
|---|---|---|---|---|---|---|---|
| ID | | | | | | | |
| XXXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | XXX | xxx | Normal/Abnormal | xxx |
| XXXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | XXX | XXX | Normal/Abnormal | xxx |
| XXXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | XXX | XXX | Normal/Abnormal | XXX |
| XXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | XXX | xxx | Normal/Abnormal | XXX |
| XXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | XXX | xxx | Normal/Abnormal | XXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# Listing 16.3.4 Listing of Patient 12-Lead electrocardiogram

| Unique | | Assessment | Date and Time of ECG | | | | |
|---|---|---|---|---|---|---|---|
| Patient ID | Visit | Done | assessment | Parameter | Result | Unit | Interpretation |
| xxxxxx | XXX | Yes/No | DD-MMM-YYYY/HH:MM | XXX | XXX | XXX | xxx |
| XXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | XXX | XXX | XXX | XXX |
| XXXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | XXX | XXX | XXX | XXX |
| XXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | XXX | XXX | XXX | XXX |
| XXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | xxx | XXX | XXX | xxx |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# Listing 16.3.5.1 Listing of Patient Haematology Parameters

| Unique | | Sample | Date and Time of | Lab | | | |
|---|---|---|---|---|---|---|---|
| Patient ID | Visit | Collected | sample collection | Parameter | Result | Unit | Interpretation |
| xxxxxx | XXX | Yes/No | DD-MMM-YYYY/HH:MM | xxx | XXX | XXX | xxx |
| XXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | XXX | XXX | XXX | XXX |
| XXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | XXX | XXX | XXX | XXX |
| XXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | XXX | XXX | XXX | XXX |
| XXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | xxx | XXX | XXX | XXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# Listing 16.3.5.2 Listing of Patient Serum Chemistry Parameters

| Unique | | Sample | Date and Time of | Lab | | | |
|---|---|---|---|---|---|---|---|
| Patient ID | Visit | Collected | sample collection | Parameter | Result | Unit | Interpretation |
| XXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | xxx | XXX | XXX | xxx |
| XXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | XXX | XXX | XXX | XXX |
| XXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | XXX | XXX | XXX | XXX |
| XXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | XXX | XXX | XXX | XXX |
| XXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | xxx | XXX | XXX | XXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# Listing 16.3.5.3 Listing of Patient Urine Routine and Microscopy Parameters

| Unique | | Sample | Date and Time of | Lab | | | |
|---|---|---|---|---|---|---|---|
| Patient ID | Visit | Collected | sample collection | Parameter | Result | Unit | Interpretation |
| XXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | xxx | XXX | XXX | xxx |
| XXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | XXX | XXX | XXX | XXX |
| XXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | XXX | XXX | XXX | XXX |
| XXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | XXX | XXX | XXX | XXX |
| XXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | xxx | XXX | XXX | XXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# Listing 16.3.5.4 Listing of Patient Thyroid Function Tests

| Unique | | Sample | Date and Time of | Lab | | | |
|---|---|---|---|---|---|---|---|
| Patient ID | Visit | Collected | sample collection | Parameter | Result | Unit | Interpretation |
| XXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | xxx | Xxx | XXX | xxx |
| XXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | XXX | Xxx | XXX | XXX |
| XXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | XXX | Xxx | XXX | XXX |
| XXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | XXX | Xxx | XXX | XXX |
| XXXXXX | XXX | Yes/No | DD-MMM-YYYY/HH:MM | xxx | Xxx | XXX | XXX |